CLINICAL TRIAL: NCT04887194
Title: A Two-cohort, Two-part, Phase 1, Multicenter, Open-label, Fixed-sequence, Drug-Drug Interaction and QTc Assessments of Sitravatinib Followed by Combination Treatment With Nivolumab in Patients With Advanced Solid Malignancies
Brief Title: PK Study to Assess Drug-drug Interaction and QTc Between Sitravatinib and a Cocktail of Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 516-010
Record Dates: First submitted 2021-05-04; First posted 2021-05-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — sitravatinib; Warfarin; Dextromethorphan; Acetylcysteine; Midazolam; Digoxin; Rosuvastatin Calcium; Nivolumab

STUDY DESIGN:
Intervention Model Description: Two Part, Phase 1 study enrolling patients with advanced tumor types into two cohorts: drug-drug interaction (DDI) and QTc. All patients receive the same anticancer treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1, Part 1: Sitravatinib monotherapy (DDI cohort) (Experimental): To evaluate the potential for drug-drug interactions (DDI) with sitravatinib monotherapy. To determine the effect of sitravatinib on the pharmacokinetics (PK) of midazolam (CYP3A4 probe substrate), warfarin (CYP2C9 probe substrate), dextromethorphan (CYP2D6 probe substrate), rosuvastatin (BCRP probe substrate), and digoxin (P-gp probe substrate).
  Interventions: Drug: Sitravatinib; Drug: Warfarin; Drug: Dextromethorphan; Drug: Midazolam; Drug: Digoxin; Drug: Rosuvastatin
- Phase 1, Part 1: Sitravatinib monotherapy (QTc cohort) (Experimental): To evaluate the QTc prolongation risk for sitravatinib in patients with advanced/metastatic solid tumors via C-QTc modeling.
  Interventions: Drug: Sitravatinib
- Phase 1, Part 2: Combination Therapy (both DDI and QTc cohorts) (Experimental): To evaluate safety and tolerability of Sitravatinib treatment with the addition of the checkpoint inhibitor nivolumab.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases
  Other Names: MGCD516
Drug: Warfarin — CYP2C9 probe substrate
  Other Names: Coumadin
  Arms: Phase 1, Part 1: Sitravatinib monotherapy (DDI cohort)
Drug: Dextromethorphan — CYP2D6 probe substrate
  Other Names: Robitussin
  Arms: Phase 1, Part 1: Sitravatinib monotherapy (DDI cohort)
Drug: Midazolam — CYP3A4 probe substrate
  Other Names: Versed
  Arms: Phase 1, Part 1: Sitravatinib monotherapy (DDI cohort)
Drug: Digoxin — P-gp probe substrate
  Other Names: LANOXICAPS
  Arms: Phase 1, Part 1: Sitravatinib monotherapy (DDI cohort)
Drug: Rosuvastatin — BCRP probe substrate
  Other Names: Crestor
  Arms: Phase 1, Part 1: Sitravatinib monotherapy (DDI cohort)
Drug: Nivolumab — Nivolumab is a programmed death receptor (PD-1) blocking antibody
  Other Names: OPDIVO
  Arms: Phase 1, Part 2: Combination Therapy (both DDI and QTc cohorts)

SUMMARY:
Study 516-010 is an open-label Phase 1, drug-drug interaction and QTc study evaluating the effect of sitravatinib on probe substrates for CYP450 enzymes and BCRP and P-gp transporters.

DETAILED DESCRIPTION:
Part 1 of this study is designed to evaluate the potential for drug-drug interactions and QTc effects with sitravatinib monotherapy when administered with probe drugs for specific cytochrome P450 (CYP) enzymes (CYP2C9, CYP2D6, and CYP3A4) and P-glycoprotein (P-gp) and breast cancer resistance protein (BCRP) transporters

Part 2 allows for patients to continue sitravatinib treatment with the addition of the checkpoint inhibitor Nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of unresectable advanced/metastatic solid tumor
* Life expectancy of at least 3 months
* Adequate bone marrow and organ function

Exclusion Criteria:

* Ongoing medical condition or need for treatment with medication that may affect the PK of study treatments during Part 1
* Immunocompromising conditions
* Impaired heart function
* Active or prior documented autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
PK parameters of probe drugs; AUC from time zero to the last data point (AUC-last) | Part 1; 1-20 Days
  (warfarin, dextromethorphan, midazolam, digoxin, and rosuvastatin) derived from the plasma concentration time profile before and after oral administration of sitravatinib
PK parameters of probe drugs; AUC from time zero to infinity (AUC∞) | Part 1; 1-20 Days
  (warfarin, dextromethorphan, midazolam, digoxin, and rosuvastatin) derived from the plasma concentration time profile before and after oral administration of sitravatinib
PK parameters of probe drugs; C-max | Part 1; 1-20 Days
  (warfarin, dextromethorphan, midazolam, digoxin, and rosuvastatin) derived from the plasma concentration time profile before and after oral administration of sitravatinib
Adverse Events | Through study completion, an average of 12 months
  Characterization of AEs by incidence, severity, timing, seriousness & relationship to study treatment

SECONDARY OUTCOMES:
Plasma PK parameters of sitravatinib and M10; C-max | 1-20 Days
  C-max
Plasma PK parameters of sitravatinib and M10; AUC over the dosing interval (AUC) | 1-20 Days
  AUC over the dosing interval (AUC)
Plasma PK parameters of sitravatinib and M10; trough plasma concentration (C-trough) | 1-20 Days
  trough plasma concentration (C-trough)
Plasma PK parameters of sitravatinib and M10; time to maximum concentration (t-max) | 1-20 Days
  time to maximum concentration (t-max)
Adverse Events | 1-20 Days
  Safety characterized by type, incidence, severity, timing, seriousness & relationship to study treatment of adverse events, and laboratory abnormalities
QT/QTc | Part 1: Pre-dose to Day 10 (QTc cohort); Part 1: Pre-dose to Day14 (DDI cohort)
  ECG data

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Chin, MD, Study Director — Mirati Therapeutics Inc.
Locations (5):
- United States (5):
  - Goshen Health, Goshen, Indiana
  - NEXT Oncology, Austin, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
  - MultiCare Health System, Tacoma, Washington